CLINICAL TRIAL: NCT06712459
Title: Integrated Molecular and Clinical Profiling of Transformed Splenic Marginal Zone Lymphoma
Status: Recruiting | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG54
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Transformed Splenic Marginal Zone Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Diagnostic tumor material collected at the time of histological transformation (mandatory), from spleen, lymph node, extra-nodal site, peripheral blood or bone marrow. If available, also SMZL diagnostic tumor material (from spleen, peripheral blood and/or bone marrow) collected at the time diagnosis will be collected (not mandatory).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Histological transformation in Splenic Marginal Zone Lymphoma (t-SMZL) represents an unmet clinical and biological need, invariably associated with poor prognosis and reduced overall survival. At the present time, there are no recommended treatments intended specifically to t-SMZL and little is known about t-SMZL genetic complexity. The aim of this study is to provide information that will help clinicians to better understand the complexity of the disease. The information gained from this study will also lead to more specific and effective treatment for patients with t-SMZL.

DETAILED DESCRIPTION:
Already existing and coded tumor biological material and health-related patient data will be retrospectively collected from institutional biobanks and patients' charts or electronic medical records upon receipt of ethical approval. Each patient enrolled in the study will be assigned a unique identification numerical code upon registration in the study. The unique identification code will be used to record health-related data and to label biological samples. Health-related data will be collected by electronic case report form (e-CRF) system. Data quality will be insured by query generation.

Annotated baseline features will include: date of diagnosis, date and tissue type of histological sample collected at diagnosis (spleen and/or bone marrow), age, gender, Eastern Cooperative Oncology Group - Performing Status (ECOG-PS), Ann Arbor stage, Lactate Dehydrogenase (LDH), number and location of extranodal sites, bone marrow involvement and percentage, peripheral blood involvement, bulky disease (>7 cm), number of nodal sites, B symptoms, hemoglobin, platelets, lymphocytes, beta-2-microglobulin, albumin, Hepatitis C Virus (HCV) infection, serum paraprotein and type.

Annotated follow-up features will include: the date of progression to a disease requiring treatment, type of first line treatment, date of start of the first line treatment, date of progression after first line treatment, date of the second line treatment, type of second line treatment.

Annotated transformation features will include: date of transformation, date and type of histological sample collected at transformation (spleen and/or bone marrow and/or lymph node and/or other site), histological transformation type and relative molecular data (if available), ECOG-PS, Ann Arbor stage, LDH, number and location of extranodal sites, bone marrow involvement and percentage, peripheral blood involvement, bulky disease (>7 cm), number of nodal sites, B symptoms, hemoglobin, platelets, lymphocytes, beta-2-microglobulin, albumin, serum paraprotein, and type.

Survival features will include the date of death, cause of death, date of last follow-up.

Mutation analysis, immunoglobulin gene rearrangement analysis, copy number aberration analysis, structural variant analysis, and DNA methylation profile will be performed by Next Generation Sequencing (NGS) of genomic DNA extracted from the biological sample available for the analysis. Gene expression will be assessed by NGS of RNA extracted from from the biological sample available for the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older, regardless of the gender;
2. Diagnosis of HT of SMZL (both at baseline, co-occurring with diagnosis of SMZL, or during the natural history of the disease);
3. Availability of diagnostic tumor material (either frozen or FFPE) from spleen, lymph node, extra nodal site, peripheral blood or bone marrow collected at the time of histological transformation. Tumor material (either frozen or FFPE), from spleen, peripheral blood or bone marrow, collected at the time of SMZL diagnosis will be also collected, if available;
4. Availability of the baseline and follow-up annotations.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with transformed SMZL
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mutations, copy number abnormalities and structural variants at SMZL diagnosis and at HT | 30 months: from the end of samples collection to the end of study analysis
Quantification and qualification of lesions acquired at the time of HT. | 30 months: from the end of samples collection to the end of study analysis
Prevalence of clonal relationship between SMZL and HT | 30 months: from the end of samples collection to the end of study analysis

SECONDARY OUTCOMES:
Prevalence of HT molecular subtypes defined by genetic lesions | 30 months: from the end of samples collection to the end of study analysis
Prevalence of Histological Transformation (HT) molecular subtypes defined by gene expression | 30 months: from the end of samples collection to the end of study analysis
Prevalence of HT molecular subtypes defined by genetic methylation profile | 30 months: from the end of samples collection to the end of study analysis
Prevalence of molecular features in relation with clinical, laboratory and radiological/Positron Emission Tomography (PET) features at SMZL diagnosis and at HT | 30 months: from the end of samples collection to the end of study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Luca Arcaini, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo; Davide Rossi, MD, Study Chair — Oncology Institute of Southern Switzerland (IOSI) and Institute of Oncology Research (IOR)
Locations (7):
- Columbia University, New York, New York, United States
- Universitz Hospitals Leuven, Leuven, Belgium
- Hôpital Saint Louis, Paris, France
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Hospital Clínic de Barcelona, Barcelona, Spain
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland
- University Hospitals Dorset, Bournemouth, United Kingdom